CLINICAL TRIAL: NCT01972412
Title: Telephone Support for Self-monitoring of Persons With Diabetes Mellitus Using the Chronic Care Model
Brief Title: Telephone Use for Care of Persons With Diabetes Mellitus.
Acronym: TCDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Tânia Alves Canata Becker, Telephone Support for self-monitoring of persons with diabetes mellitus, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EERP - 146.171
Record Dates: First submitted 2013-03-26; First posted 2013-10-30 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Diabetes Mellitus
Keywords: nursing care; diabetes mellitus; phone support; chronic care model
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telephone support (Other): Intervention type: Telephone support for four months.
  Interventions: Behavioral: telephone support

INTERVENTIONS:
Behavioral: telephone support — Telephone support for four months about healthy diet, physical activity and medication use.

SUMMARY:
The purpose of this study is to determine whether phone use contributes to diabetes control.

DETAILED DESCRIPTION:
Studies reinforce the need to test innovative care that can serve more patients, since education is a key element for the accession to the treatment of diabetes. Recently, an innovative, feasible and low cost presented in the literature is the use of telephone support as an intervention strategy This study aims to evaluate the implementation of a telephone support for self-monitoring of people with diabetes mellitus treated in ribeirão Preto.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus type 2
* age
* ability to listen and answer questions

Exclusion Criteria:

* often present less than 75% participation in the proposed activities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-01 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Telephone Support for self-monitoring of persons with diabetes mellitus using the Chronic Care Model | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Tânia A Canata Becker, Master, Principal Investigator — University of São Paulo at Ribeirão Preto College of Nursing
Locations (2):
- Brazil (2):
  - University of São Paulo at Ribeirão Preto College of Nursing, Ribeirão Preto, São Paulo
  - Universidade de São Paulo, Ribeirão Preto, São Paulo

REFERENCES:
- [Derived] Becker TAC, Teixeira CRS, Zanetti ML, Pace AE, Almeida FA, Torquato MTDCG. Effects of supportive telephone counseling in the metabolic control of elderly people with diabetes mellitus. Rev Bras Enferm. 2017 Jul-Aug;70(4):704-710. doi: 10.1590/0034-7167-2017-0089. English, Portuguese. PMID 28793098
- See also: Affiliated to the International Diabetes Federation. — http://www.diabetes.org.br/